CLINICAL TRIAL: NCT06857708
Title: The Management of Necrotizing Soft Tissue Infection Wounds With Cytal® Wound Matrix and MicroMatrix®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin T. Miller (Other)
Responsible Party: Sponsor-Investigator, Benjamin T. Miller, Assistant Professor of Surgery, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 23-1221
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Necrotizing Fascitis; Necrotizing Soft Tissue Infection
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interventional arm (Experimental): This arm will receive application of Cytal® Wound Matrix and MicroMatrix®
  Interventions: Device: Cytal® Wound Matrix; Device: MicroMatrix®
- Standard of Care Arm (No Intervention)

INTERVENTIONS:
Device: Cytal® Wound Matrix — This is the only study to use this intervention in necrotizing soft tissue wounds
  Arms: Interventional arm
Device: MicroMatrix® — This is the only study to use this intervention in necrotizing soft tissue wounds
  Arms: Interventional arm

SUMMARY:
This is a prospective, pilot, parallel group, randomized controlled trial with 1:1 allocation. This will be a single center study coordinated at the Cleveland Clinic Foundation (CCF) Main Campus in Cleveland, Ohio. Data will be collected in a secure manner using REDCap housed at CCF. The study will consist of 2 arms: treatment with Cytal® Wound Matrix 2-Layer and MicroMatrix® (Integra LifeSciences, Plainsboro Township, NJ, U.S.A.) versus standard of care dressings. Wound debridement procedures will be performed by surgical staff at CCF. A co-investigator trained in the application of Cytal® Wound Matrix and MicroMatrix® will apply these treatments as outlined in section 6.1.2 Administration. This study will be conducted with IRB approval and written informed consent of each participant enrolled. The trial will be registered at ClinicalTrials.gov before the first participant is enrolled.

DETAILED DESCRIPTION:
Necrotizing fasciitis (NF) is a type of soft tissue infection that is characterized by necrosis of the subcutaneous tissues and muscle fascia. Prompt diagnosis and surgical exploration are crucial in the management of these potentially fatal infections.1,2 For most patients, this requires an initial extensive, wide debridement with repeated inspection and debridement every 24-48 hours to remove all necrotic tissue.3 As a result, tissue reconstruction often necessitates flap surgery with autologous, split-thickness skin grafting (STSG) for sufficient coverage. The process during which the wound bed becomes ready for skin grafting can be lengthy, arduous, and often times costly. Post-discharge regimens may consist of pain management for daily dressing changes, nutritional supplements, multiple follow up visits in clinic and likely the involvement of a plastic and reconstructive surgeon.4 Therefore, strategies to promote the healing of these wounds may significantly improve the morbidity of this disease.

One such adjunct to the management of wounds is the use of mammalian-derived extracellular matrices (ECM). Multiple published case reports have demonstrated the safety and efficacy of ECM in the healing process of complex wounds.5-12 A randomized controlled trial was conducted in patients with chronic venous ulcers using an ECM derived from the submucosal layers of the porcine jejunum.8 Their findings demonstrated significant improvement in wound healing as compared to a standard-care group at 12 weeks of treatment (55% vs 34%, p = 0.196).

Cytal® and MicroMatrix® (Integra LifeSciences, Plainsboro Township, NJ, U.S.A.) are acellular, ECM products derived from porcine bladder epithelial basement membrane and tunica propria. It is thought that these products provide an optimal environment for healing by providing a scaffold for tissue regeneration and promoting neovascularization. These products have previously been demonstrated to improve healing in NF wounds.9-12 However, to date, there have been no randomized controlled trials evaluating the efficacy of ECM in the healing of NF wounds. We hypothesize that wound beds treated with Cytal® and MicroMatrix® will have a significantly decreased time to skin graft readiness as compared to those treated with standard of care wound management.

This is a prospective, pilot, parallel group, randomized controlled trial with 1:1 allocation. This will be a single center study coordinated at the Cleveland Clinic Foundation (CCF) Main Campus in Cleveland, Ohio. Data will be collected in a secure manner using REDCap housed at CCF. The study will consist of 2 arms: treatment with Cytal® Wound Matrix 2-Layer and MicroMatrix® (Integra LifeSciences, Plainsboro Township, NJ, U.S.A.) versus standard of care dressings. Wound debridement procedures will be performed by surgical staff at CCF. A co-investigator trained in the application of Cytal® Wound Matrix and MicroMatrix® will apply these treatments as outlined in section 6.1.2 Administration. This study will be conducted with IRB approval and written informed consent of each participant enrolled. The trial will be registered at ClinicalTrials.gov before the first participant is enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years) with a diagnosis of necrotizing fasciitis
2. Wound ≥ 30 cm2
3. The participant is willing and able to adhere to protocol requirements and agrees to participate in the study program and comply with the study follow-up regimen.

Exclusion Criteria:

1. Burn as etiology of wound
2. Acute osteomyelitis requiring active treatment
3. Known allergy, hypersensitivity, or objection to porcine materials
4. Pregnant participants
5. Lack of English language fluency
6. Participant report of concurrent participation in another clinical trial that would interfere with this study
7. Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to readiness for grafting of the wound bed | From randomization to readiness for grating, up to 12 weeks

SECONDARY OUTCOMES:
Relative wound healing as assessed by the Photographic Wound Assessment Tool (PWAT) | From randomization to readiness for grating, up to 12 weeks
  Relative wound healing as assessed by the Photographic Wound Assessment Tool (PWAT) between the two study arms
Assess the relative rate of wound infection, seroma, hematoma, and need for re-intervention (including incision and drainage) | From randomization to readiness for grating, up to 12 weeks
  To assess the relative rate of wound infection, seroma, hematoma, and need for re-intervention (including incision and drainage) between the treated and untreated wound beds
To assess the rate of product excision resulting from wound complications, allergic reaction, or intolerance to the product | From randomization to readiness for grating, up to 12 weeks
To assess relative rates of wound closure, measured as the proportion of the remaining wound area compared to the starting wound area | From randomization to readiness for grating, up to 12 weeks
To assess relative skin graft size as a percentage of starting wound area | From randomization to readiness for grating, up to 12 weeks
To assess the relative percentages of skin graft take | From randomization to readiness for grating, up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States